CLINICAL TRIAL: NCT03878732
Title: Bindex for Osteoporosis Diagnostics
Status: Completed | Type: Observational
Sponsor: Bone Index Finland Ltd (Industry)
Collaborators: New Mexico Clincial Research & Osteoporosis Center, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Bind2301
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Caucasian female
  Interventions: Diagnostic Test: Bindex measurement
- Hispanic female
  Interventions: Diagnostic Test: Bindex measurement

INTERVENTIONS:
Diagnostic Test: Bindex measurement — One time bone density measurement with ultrasound device

SUMMARY:
Osteoporosis is a disease that leads to impaired skeletal strength and increased fracture risk. Among 200 million osteoporotic patients most are diagnosed only after several fractures. Furthermore, the progressively aging population will increase the prevalence of osteoporosis. It is estimated that over 75% of osteoporotic patients are not diagnosed and does not receive treatment for their condition. Bindex ultrasound device has been developed and validated in Caucasian female population. In this study, diagnostic thresholds for density index as determined with Bindex will be evaluated in two different ethnic populations.

DETAILED DESCRIPTION:
Currently, the diagnosis of osteoporosis is based on the measurement of bone mineral density (BMD), using axial dual energy X-ray absorptiometry (DXA) of the hip and/or the lumbar spine at special healthcare.

Application of diagnostic thresholds determined against BMD have been suggested by International Society for Clinical Densitometry (ISCD) for use with peripheral bone densitometry devices (90% sensitivity and 90% specificity). These thresholds have been determined and validated for Bindex in Caucasian female population.

This study focuses on clinical validation of the ultrasound device (Bindex®, Bone Index Finland Ltd., www.boneindex.com) device and Density Index (DI), a diagnostic parameter reported by Bindex. The predetermined thresholds for DI will be evaluated by measuring 70 osteoporotic and 70 healthy patients with Bindex and DXA in each selected patient groups. The feasibility of DI for diagnostics of osteoporosis in these groups will be assessed.

ELIGIBILITY:
Inclusion Criteria for all:

* Postmenopausal status
* Age at 50 years or over
* Caucasian or Hispanic race (number shall be controlled, 140 in each group)
* Body mass index (BMI < 35)

Additional criteria for Osteoporotic group

- T-Score (NHANES database) -2.5 or lower at femoral neck or total femur

Additional criteria for non-osteoporotic group

- T-Score (NHANES database) > -2.5 at femoral neck or total femur

Exclusion Criteria:

for non-osteoporotic groups (Hispanic or Caucasian)

* Previous osteoporosis diagnosis
* Previous or current use of anti-fracture medication

Ages: 50 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Review history. No genetic testing shall be done or confirmation of external sexual organs.Transgender individuals will not be included in the study population.
Study Population: Random sample of eligible female subjects who are being treated at collaborating clinic.
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of DI | 3/11/2019-11/29/2019
  Sensitivity and specificity of DI in caucasian and hispanic groups

CONTACTS AND LOCATIONS:
Overall Officials: Janne Karjalainen, Study Chair — Bone Index Finland Ltd
Locations (1):
- New Mexico Clincial Research & Osteoporosis Center, Inc., Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No